CLINICAL TRIAL: NCT04282031
Title: A Phase 1/2a Study to Evaluate the Tolerability, Safety, Pharmacokinetics and Efficacy of BPI-1178 Alone in Advanced Solid Tumor and of BPI-1178 in Combination With Endocrine Therapy in Advanced HR+/HER2- Breast Cancer
Brief Title: A Study of BPI-1178 in Patients With Advanced Solid Tumor and HR+/HER2- Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beta Pharma (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BPI-1178-2019-001
Record Dates: First submitted 2020-02-18; First posted 2020-02-24 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Advanced Solid Tumor; HR+/HER2- Breast Cancer
MeSH Terms: interventions — Fulvestrant; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- phase 1 (dose escalation study, dose expansion study and PK trail) (Experimental): Participants will first receive single dose BPI-1178 orally at dose levels of 25mg, 75mg, 150mg, 250mg, 400mg and 500mg followed by a 7-day washout period , and then start receiving the 28 days/cycle continuous treatment until disease progression or unacceptable toxicity. After the 500 mg dose escalation trial is completed, the PK study will be conducted for the 400 mg dose group, the 300 mg dose group and the 200 mg dose group.
  Interventions: Drug: BPI-1178
- phase 2a cohort A (Experimental): Participants will receive BPI-1178 at dose levels of MTD, MTD-1 or MTD-2 in combination with fulvestrant for 3 consecutive weeks, followed by 1 week drug withdrawal or continuous dosing for 28 days, in each 28-day treatment cycle, until disease progression or unacceptable toxicity.
  Interventions: Drug: BPI-1178; Drug: Fulvestrant
- phase 2a cohort B (Experimental): Participants will receive BPI-1178 at dose levels of MTD, MTD-1 or MTD-2 in combination with letrozole for 3 consecutive weeks, followed by 1 week drug withdrawal or continuous dosing for 28 days, in each 28-day treatment cycle, until disease progression or unacceptable toxicity.
  Interventions: Drug: BPI-1178; Drug: Letrozole

INTERVENTIONS:
Drug: BPI-1178 — BPI-1178 once daily on Days 1 to 21 of a 28-day cycle
Drug: Fulvestrant — Fulvestrant 500mg intramuscularly on Days 1 and 15 of Cycle 1, and on Day 1 of Cycle 2 and beyond
  Arms: phase 2a cohort A
Drug: Letrozole — Letrozole 2.5 mg once daily of a 28-day cycle
  Arms: phase 2a cohort B
Drug: BPI-1178 — BPI-1178 once daily of a 28-day cycle
  Arms: phase 2a cohort A; phase 2a cohort B

SUMMARY:
BPI-1178 is a novel, orally administered inhibitor of both cyclin-dependent kinase 4（CDK4）and CDK6 kinase activity. This Phase I study is a first-in-human (FIH) clinical trial designed to evaluate the safety, tolerability, and pharmacokinetic (PK) profile of oral BPI-1178 in patients with advanced solid tumors. The Phase IIa trial is designed to investigate the anti-tumor activity and safety of BPI-1178 in combination with endocrine therapy in patients with HR+/HER2-advanced breast cancer and to determine the dosing regimen for combination with endocrine therapy in a later confirmatory study.

DETAILED DESCRIPTION:
This is a study which consists of phase １study（dose-escalation study、dose-expansion study and PK trial） and phase 2a study.

Phase 1 study will adopt the classical 3+3 dose escalation design, exploring the safety and tolerance of 6 dose cohorts (25mg, 75mg, 150mg, 250mg, 400mg and 500mg) in subjects with advanced solid tumor and determining the maximum tolerated dose of BPI-1178 for phase 2a study.

Phase 2a is an open-label clinical study in subjects of HR+/HER2- breast cancer using 3+3 design, to evaluate the efficacy and safety of BPI-1178 in combination with endocrine therapy. Cohort A is BPI-1178 in combination with fulvestrant for advanced or recurrent HR+/HER2- breast cancer after failure or intolerance of non-fulvestrant first-line endocrine therapy. Cohort B is BPI-1178 in combination with letrozole for advanced or relapse more than 1 year after the end of adjuvant endocrine therapy as first-line treatment.

Phase 1 and 2a consist of screening period (28 days before enrollment), treatment period and follow up period (every 3 months until death or the end of study). Phase 1 study: Subjects in each dose group will first receive a single dose. After a single dose for washout period, if the subject has no dose-limiting toxicity (DLT) related to the investigational product, the subject will enter the continuous dose cycle and receive continuous dose in a 28-day treatment cycle (single daily dose for 3 consecutive weeks/drug withdrawal for 1 week) .Once the maximum tolerated dose (MTD) is reached in phase 1, phase 2a study will explore the dose of BPI-1178 from MTD in combination with fulvestrant or letrozole. Phase 2a study: Subjects in Cohort A and Cohort B with intermittent dosing (3-week continuous dosing followed by 1-week rest) and continuous dosing (28-day continuous dosing) will be received in combination with fulvestrant or letrozole. Each 28-day is a complete treatment cycle during the concomitant-drug period.

Dose limiting toxicity (DLT) will be recorded for the single dose period of 7 days and the multiple dose period up to 28 days in phase 1 study, as well as 28 days after the first dose of BPI-1178 in phase 2a. Efficacy will be evaluated by RECIST v1.1 and the Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) every 2 months. Adverse events will be monitored throughout the trial. Other exploration of pharmacokinetic information will be assessed throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent prior to any study specific procedures.
2. Male or female, aged ≥18 years.
3. Subjects with advanced solid tumors:

   * Phase 1: Histologically or cytologically confirmed, locally advanced (not amenable to curative treatment of surgical resection or radiation therapy), recurrent, or metastatic solid tumors that were refractory to standard therapy or for which no standard-of-care therapy.
   * Phase 2a Cohort A: HR+/HER2- locally advanced, recurrent, or metastatic breast cancer with disease progression after first-line endocrine therapy (not fulvestrant) or intolerant of it, histologically confirmed by the primary and/or metastatic lesions, not amenable to chemotherapy or curative treatment of surgical resection or radiation therapy; if the pathology of the primary and metastatic lesions are inconsistent, diagnosis should be based on metastatic lesions' pathology.
   * Phase 2a Cohort B: HR+/HER2- locally advanced, recurrent, or metastatic breast cancer with no prior systemic therapy in this disease setting or relapse more than 1 years from completion of adjuvant endocrine therapy, histologically confirmed by the primary and/or metastatic lesions, not amenable to chemotherapy or curative treatment of surgical resection or radiation therapy; if the pathology of the primary and metastatic lesions are inconsistent, diagnosis should be based on metastatic lesions' pathology.
   * Female patients with breast cancer at Phase IIa must also meet the following criteria:

     (1) Postmenopausal patients must meet at least one of the following criteria:
     1. Age ≥ 60 years old;
     2. Patients < 60 years of age who have menstruation ceased for at least 12 consecutive months and have not received chemotherapy, tamoxifen, toremifene or ovarian function inhibitors, and have blood estrogen and FSH levels within the reference range for postmenopausal women;
     3. Previous bilateral ovariectomy;
     4. Patients < 60 years of age who are being treated with tamoxifen or toremifene with blood estrogen and FSH levels within the reference range for postmenopausal women.

     (2) Premenopausal/perimenopausal patients must meet the following criteria: Premenopausal/perimenopausal patients requiring ovarian function suppression must start treatment at least 4 weeks prior to enrollment and the treatment should be maintained during the trial.
4. At least 1 measurable lesion based on the RECIST v1.1 criteria.
5. Life expectancy≥ 12 weeks.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS)≤1.
7. Adequate bone marrow and organ function, defined as following:

   1. absolute neutrophil count≥1.5×10^9/L, platelets≥100×10^9/L, hemoglobin≥100 g/L;
   2. total bilirubin≤1.5×ULN(≤3×ULN for Gilbert syndrome), alanine aminotransferase and aspartate aminotransferase≤3×ULN;
   3. serum creatinine≤1.5×ULN or a creatinine clearance calculated by Cockcroft-Gault formula≥50 mL/min; urinary protein measured by semi-quantitative method<2+; if urinary protein measured by semi-quantitative method at baseline ≥2+, 24-h urinary protein<1g;
   4. activated partial thromboplastin time and international normalized ratio≤1.5×ULN;
   5. LVEF≥50%;
   6. Corrected QT interval (QTcF)<450ms for men and <470ms for women at resting.
8. Female subjects should take effective contraceptive methods during the study and for 60 days after the last dose of BPI-1178, and must have a negative pregnancy test prior to dosing if of child-bearing potential, or must have evidence of non-child-bearing potential; male subjects should take effective contraceptive methods during the study and for 120 days after the last dose of BPI-1178.
9. All subjects must have enough mental behavior ability, understand the nature and significance of the study, as well as the risks associated with the study.

Exclusion Criteria:

1. Currently receiving or have received any CDK4/6 inhibitors.
2. Have had allergies or history of severe allergies.
3. Have participated in any clinical trials within 4 weeks prior to the dosing of BPI-1178.
4. Have received anti-tumor therapy (including chemotherapy, endocrine therapy, targeted therapy, immunotherapy, tumor embolization, etc.; have received radiotherapy within 2 weeks before taking the investigational product) within 4 weeks before starting to take the investigational product <except for premenopausal/perimenopausal patients with Gonadotropin-releasing hormone analogues [GnRHa] therapy allowed in Phase IIa study>.
5. Other malignancies present or previously present at the time of enrollment or still under treatment at the time of enrollment (only applicable to Phase IIa study)
6. Any toxicity related to previous treatment before enrollment defined by CTCAE (v5.0) Grade≥2 (except hair loss).
7. Presence of third interstitial fluid that cannot be controlled by drainage or other methods (such as large amounts of pleural fluid and ascites).
8. Requiring long-term treatment of steroid.
9. Having uncorrectable hypokalemia and hypomagnesemia at enrollment.
10. Meet any of the following criteria: Various clinically significant heart rhythm and conduction abnormalities, such as atrial fibrillation, complete left bundle branch block, Level III conduction block, Level II conduction block, and PR interval > 250 msec; Various factors that might increase risks of QT increased or arrhythmia events, e.g., symptomatic cardiac failure - New York Heart Association (NYHA) class 2-4, long QT syndrome congenital, Brugada syndrome, previous histories of QT increased (> 470 ms for males, > 480 ms for females) or TdP attack, first degree relative of the family with long QT syndrome or sudden death before 40 years' old with unexplained cause, and concomitant medication which may prolong QT interval; Suffering from following diseases within 6 months prior to administration of investigational product, including unstable angina pectoris, myocardial infarction, coronary heart disease, cerebrovascular accident or pulmonary embolism, or accepting cardiac revascularization.
11. Known active infection, such as hepatitis B (HBV DNA ≥ 200 IU/mL), hepatitis C, human immunodeficiency virus (HIV) infection.
12. Have a history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
13. Based on the judgement of investigators, there might be multiple factors which could impact taking and absorption of BPI-1178, including gastrointestinal factors (e.g., obviously uncontrollable inflammatory gastrointestinal disorder, abdominal colostomy within 6 months or previous history of gastrointestinal perforation, extensive resection of small intestine and requirement of tube feeding or water/ nutritional supplement by parenteral route, inability to swallow, chronic diarrhoea and intestinal obstruction, etc.)
14. Have spinal cord compression, metastases of the meninges, or brain metastases with obvious symptoms. The following cases of brain metastases without symptoms can be enrolled: brain metastases without obvious symptoms diagnosed at screening visit, steroids and/or local treatment not required judged by investigator; brain metastases without obvious symptoms after local treatment (such as radiotherapy), and steroids and/or antiepileptic therapy has stopped for at least 7 days before the first dosing of BPI-1178.
15. In the judgment of the investigator, have a concomitant disease (such as severe hypertension, diabetes, thyroid disease, severe infection, portal hypertension, cirrhosis, etc.) that would endanger the subjects' safety or affect the completion of the study.
16. Have had major surgery (craniotomy, thoracotomy, or laparotomy) or unhealed wounds, ulcers, or fractures within 4 weeks prior to the dosing of BPI-1178.
17. Pregnant or lactating women, or fertile women with pregnancy test positive at baseline.
18. Any factors that may endanger subject's safety and may affect subject's compliance with the study.
19. Drug abuse, alcoholic addiction, medical and mental illness and social barriers judged by investigator, which may interfere the subjects' participation in the study or affect the evaluation of study endpoints . Any factor that investigator believes may make the subjects not suitable to receive BPI-1178. Subjects are unwilling or unable to comply with the requirements of the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
phase 1 and 2a: Number of subjects with dose limiting toxicity (DLT) | Up to Day 28 of Cycle 1 (28 days/cycle)
phase 1: Maximum tolerated dose (MTD) | Up to Day 28 in Cycle 1 (28 days/cycle)
phase 2a: Objective response rate (ORR) | Up to approximately 18 months

SECONDARY OUTCOMES:
phase 1 and 2a: Number of subjects with adverse events | Up to 30 days after the last dose of BPI-1178
phase 1: Objective response rate (ORR) | Up to approximately 18 months
Phase 1 and 2a: Maximum plasma concentration (Cmax) of BPI-1178 and its main metabolites | From single dosing in phase 1 or from baseline in phase 2a to the end of Cycle 1 (28 days/cycle)
Phase 1 and 2a: Peak Plasma Time (Tmax) of BPI-1178 and its main metabolites | From single dosing in phase 1 or from baseline in phase 2a to the end of Cycle 1 (28 days/cycle)
Phase 1 and 2a: Area under the plasma concentration versus time curve (AUC) of BPI-1178 and its main metabolites | From single dosing in phase 1 or from baseline in phase 2a to the end of Cycle 1 (28 days/cycle)

OTHER OUTCOMES:
Clearance of BPI-1178 and its main metabolites | From single dosing in phase 1 or from baseline in phase 2a to the end of Cycle 1 (28 days/cycle)
Half life of BPI-1178 and its main metabolites | From single dosing in phase 1 or from baseline in phase 2a to the end of Cycle 1 (28 days/cycle)
Disease control rate ( DCR) | Up to approximately 18 months
Duration of response ( DoR) | Up to approximately 18 months
Progression free survival (PFS) | Up to approximately 18 months
Overall survival (OS) | Baseline to date of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China